CLINICAL TRIAL: NCT01674608
Title: TEAM: An Multi-centre Observational Study of Early Activity and Mobilization in Australia and New Zealand
Brief Title: TEAM: Trial of Early Activity and Mobilization
Acronym: TEAM
Status: Completed | Type: Observational
Sponsor: Australian and New Zealand Intensive Care Research Centre (Other)
Collaborators: Intensive Care Foundation, Australia (Unknown)
Responsible Party: Sponsor
Other Study IDs: ICF
Record Dates: First submitted 2012-08-14; First posted 2012-08-29 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Critically Ill Adults Ventilated >24 Hours in Intensive Care
Keywords: intensive care; mobilization; rehabilitation; critical care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients in the Intensive Care Unit (ICU) traditionally receive bed rest as part of their care. They develop muscle weakness even after only a few days of mechanical ventilation that may prolong their time in ICU and in hospital, but the nature of such weakness is poorly understood.

The weakness that develops in ICU is more substantial than that which would result from bed rest alone and is referred to as ICU acquired weakness (ICUAW). This weakness might be due to the combination of inflammation and immobility. The exact mechanisms leading to the nerve and muscle damage which occurs in critical illness are not yet fully understood and require further investigation. However, it is known that ICUAW has an effect on a patient's ability to breathe without a ventilator, walk and perform simple activities (like washing and toileting) and often results in longer mechanical ventilation time and hence, longer hospital stays than might otherwise be expected. It may also affect a patient's ability to return home after their hospital stay. The recovery period in Australian and New Zealand ICU patients is unknown but a trial from Canada has reported ongoing weakness five years after leaving ICU. Weakness in survivors of intensive care is known to be a substantial problem. It is currently not known whether ICUAW may be avoided or its severity reduced with simple strategies of early exercise in ICU.

There are no data about the level of activity and mobility in critically ill patients in Australian and New Zealand ICUs. These data are urgently required to plan a program of research to test whether increasing the level of mobility and activity in our critically ill patients is safe, feasible and efficacious in terms of reducing the severity of ICUAW and improving patient-centred outcomes. The program of research will first include a study to observe the mobility levels in 25 ICUs across Australia and New Zealand to determine safety, barriers to mobility and what type of activities are undertaken by our patients.

From the observational data we plan to develop a pilot randomised controlled trial of early mobility and activity in intensive care units across Australia and New Zealand. This simple, cost-effective strategy may improve functional ability, decrease time on mechanical ventilation and improve long term outcomes in this patient group. By initiating such a program, ANZ investigators might be able to change future patient outcomes worldwide.

ELIGIBILITY:
Inclusion Criteria:

* they have received invasive mechanical ventilation for at least 24 hours, and have been in ICU less than 72 hours
* the treating clinician expects the patient to still be receiving invasive mechanical ventilation in the ICU the day after tomorrow.

Exclusion Criteria:

* Age less than 18 years old

  * Patient has a proven or suspected acute primary brain process that is likely to result in global impairment of conscious level or cognition, such as traumatic brain injury, intracranial haemorrhage, stroke, or hypoxic brain injury after cardiac arrest or asphyxiation.
  * Second or subsequent admission to ICU during a single hospital admission
  * Patient does not speak English
  * Patient has proven or suspected primary myopathic or neurological process associated with prolonged weakness, such as Guillain-Barre syndrome
  * Death is deemed imminent and inevitable
  * Inability to walk without assistance prior to the acute illness that is associated with admission to ICU (use of a cane or walker not an exclusion)
  * Cognitive impairment prior to the acute illness that is associated with admission to ICU (refer data dictionary)
  * Any written "Rest In Bed" or non-weight bearing medical order such as may occur with hip fracture, unstable spine or pelvis, pathological fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensive care unit patients
Sampling Method: Non-Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2012-07; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Best level of activity in ICU | ICU stay (average 7 days)
  Highest level of activity (11 point scale) including:
  unknown nothing (lying in bed, passive stretches) sitting in bed, active exercises in bed moved to chair (via hoist, slide etc but no standing) sitting over edge of bed standing transferring bed to chair marching on spot (at bedside) walking with assistance of 2 or more people walking with assistance of 1 person walking independently with a gait aid walking independently without a gait aid
Dosage of the best level of activity | Intensive care unit stay (average 7 days)
  The time spent performing the best level of activity and the number of times it is achieved
Time to standing in ICU | Intensive care stay (average 7 days)
  The number of days in ICU before a patient can stand

SECONDARY OUTCOMES:
Best level of activity at hospital discharge | Hospital stay (median days 14)
  Highest level of activity (11 point scale) including:
  unknown nothing (lying in bed, passive stretches) sitting in bed, active exercises in bed passively moved to chair (pat slide, hoist but no standing) sitting over edge of bed standing transferring bed to chair marching on spot (at bedside) walking with assistance of 2 or more people walking with assistance of 1 person walking independently with a gait aid walking independently without a gait aid
Time to first sit out of bed | ICU stay (average 7 days)
  The number of days until the patient can sit out of bed
Barriers to mobilisation | Intensive care unit stay (average 7 days)
  Factors that may have been a barrier to mobilizing patients in the ICU
Mobilization related adverse events | Intensive care unit stay (average 7 days)
  Adverse events that occured during patient mobilization such as an unplanned extubation or a fall to the floor
Time to first physiotherapy | Intensive care unit stay (average 7 days)
  The number of days in intensive care before the patient was reviewed by a physiotherapist
Mechanical ventilation free days | 28 days
  The number of mechanical ventilation free days to day 28
Intensive care unit free days | Day 28
  The number of days the patient spent out of ICU to day 28 (if dead = 0)
90 day mortality | 90 days
  The mortality at day 90
Health related quality of life at 6 months | 6 months
  Health related quality of life reported via telephone interview at 6 months using the EuroQoL EQ5D

CONTACTS AND LOCATIONS:
Overall Officials: Carol Hodgson, PhD, Study Chair — ANZIC-RC; Steve Webb, MD, Study Director — ANZICS CTG; Rinaldo Bellomo, MD, Study Director — ANZIC-RC; Megan Harrold, PhD Candidate, Principal Investigator — Royal Perth Hospital; Susan Berney, PhD, Principal Investigator — Austin Health; Heidi Buhr, RN, Principal Investigator — Royal Prince Alfred Hospital, Sydney, Australia; Manoj Saxena, MD, Principal Investigator — St George Hospital; Paul Young, MD, Principal Investigator — Wellington Hospital; Oystein Tronstad, PT, Principal Investigator — Prince Charles Hospital; Neil Orford, MD, Principal Investigator — Barwon Health
Locations (2):
- The Alfred, Melbourne, Victoria, Australia
- Wellington hospital, Wellington, New Zealand

REFERENCES:
- [Result] TEAM Study Investigators; Hodgson C, Bellomo R, Berney S, Bailey M, Buhr H, Denehy L, Harrold M, Higgins A, Presneill J, Saxena M, Skinner E, Young P, Webb S. Early mobilization and recovery in mechanically ventilated patients in the ICU: a bi-national, multi-centre, prospective cohort study. Crit Care. 2015 Feb 26;19(1):81. doi: 10.1186/s13054-015-0765-4. PMID 25715872
- [Derived] Tipping CJ, Bailey MJ, Bellomo R, Berney S, Buhr H, Denehy L, Harrold M, Holland A, Higgins AM, Iwashyna TJ, Needham D, Presneill J, Saxena M, Skinner EH, Webb S, Young P, Zanni J, Hodgson CL. The ICU Mobility Scale Has Construct and Predictive Validity and Is Responsive. A Multicenter Observational Study. Ann Am Thorac Soc. 2016 Jun;13(6):887-93. doi: 10.1513/AnnalsATS.201510-717OC. PMID 27015233